CLINICAL TRIAL: NCT03189446
Title: Phase II Trial of Vaginal Cuff Brachytherapy Followed by Adjuvant Chemotherapy With Carboplatin and Dose Dense Paclitaxel in Patients With High-Risk Endometrial Cancer
Brief Title: Vaginal Cuff Brachytherapy Followed by Chemotherapy in Endometrial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7964
Record Dates: First submitted 2017-05-24; First posted 2017-06-16 (Actual); Results first posted 2021-01-12 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Endometrial Cancer; Papillary Serous; Clear Cell Endometrial Cancer
Keywords: Endometrial Cancer; Gynecologic Cancer; radiation therapy
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vaginal Cuff Brachytherapy + Chemotherapy (Experimental): Vaginal cuff brachytherapy followed by Carboplatin (AUC 6) on day 1and Paclitaxel 80 mg/m2 IV over 1 hour days 1, 8, and 15 X 3 total cycles
  Interventions: Radiation: Vaginal Cuff Brachytherapy; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Radiation: Vaginal Cuff Brachytherapy — Within 12 weeks of surgery. Either LDR or HDR brachytherapy will be permitted
Drug: Carboplatin — Carboplatin IV on day 1 of a 21 day cycle for 3 cycles
Drug: Paclitaxel — Paclitaxel IV on days 1,8 and 15 of a 21 day cycle for 3 cycles

SUMMARY:
The purpose of this study is to determine the feasibility of treatment in patients with high risk endometrial cancer treated by vaginal cuff brachytherapy followed by 3 cycles of dose dense paclitaxel and carboplatin chemotherapy.

DETAILED DESCRIPTION:
Before the patient begins the study:

Endometrial cancer is commonly treated with surgery. The patient must have already had surgery including hysterectomy (removal of the uterus) prior to being considered eligible for this study. The surgery may also include removal of pelvic and para-aortic lymph nodes. Following the surgery, the doctor will identify if the patient has factors related to the cancer which places the patient at a greater risk for the cancer returning.

Prior to participating in this study there are exams, tests or procedures to find out if the patient can be treated in the study. Most are part of regular cancer care.

Treatment:

All patients will receive radiation therapy followed by three cycles of dose dense paclitaxel and carboplatin chemotherapy. Radiation therapy will be delivered either by LDR or HDR brachytherapy and must be specified at the time of enrollment. The vaginal brachytherapy should be started within 12 weeks of surgery (within 2 weeks of enrollment). Chemotherapy should start within 3 weeks of initiating brachytherapy.

Study participation will be up to two years.

ELIGIBILITY:
Inclusion Criteria:

1. All patients must have undergone hysterectomy. Bilateral salpingooophorectomy is strongly encouraged but not mandatory.
2. Pelvic and para-aortic lymphadenectomy are optional, but strongly encouraged. Peritoneal washing are optional.
3. If either a bilateral salpingo-oophorectomy or nodal dissection was not performed, post-operative pre-treatment CT/MRI is required and must not demonstrate evidence suggestive of metastatic disease (adnexa, nodes, intraperitoneal disease). Post-operative, pre-treatment CT/MRI must be performed if a pelvic and para-aortic nodal dissection was not performed.
4. All patients will be staged according to the FIGO 2009 staging system and with endometrial carcinoma (endometrioid types) confined to the corpus uteri or with endocervical glandular involvement fitting one of the following high-intermediate risk factor categories:

   * age ≥18 years with 3 risk factors
   * Risk factors:

     1. Grade 2 or 3 tumor, (+) lymphovascular space invasion, outer ½ myometrial invasion. Patients with these risk criteria may be enrolled with either positive or negative cytology.
     2. Patients with Stage II endometrial carcinoma (any histology) with cervical stromal invasion. (occult or gross involvement), with or without high-intermediate risk factors.
     3. Patients with serous or clear cell histology (with or without other high-intermediate risk factors) are eligible provided the disease is uterine-confined (with or without cervical stromal invasion or endocervical glandular involvement).
5. Patients must have GOG performance status 0, 1, or 2.
6. Patients must have adequate bone marrow, renal, hepatic and neurologic function per protocol.
7. Patients who have met the pre-entry requirements specified in protocol; testing values/results must meet eligibility criteria specified in protocol.
8. Patients must have signed an approved informed consent and authorization permitting release of personal health information.

Exclusion Criteria:

1. Patients with recurrent disease.
2. Patients with GOG performance status of 3 or 4.
3. Greater than 12 weeks elapsed from surgery to enrollment.
4. Patients have prior pelvic or abdominal radiation therapy.
5. Known hypersensitivity to any component of study treatment that resulted in drug discontinuation.
6. Significant intercurrent illness including, but not limited to, unstable angina pectoris, and cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
7. Active pregnancy or lactation.
8. Prior malignancy requiring treatment within the last 3 years.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2021-10-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Moore, MD, Principal Investigator — Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at a single institution from October 2017 to July 2019. The first patient was enrolled on October 2, 2017 and the last patient was enrolled on July 23, 2019
Pre-assignment Details: Of 39 enrolled participants, 32 met inclusion criteria and evaluable then assign to the single arm treatment.
Period: Overall Study
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Started | 32
Completed | 27
Not Completed | 5
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 64.5 [41 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 32
Body Mass Index [Median (Full Range); unit: kg/m^2] | 35.1 [24 to 68.9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Completing the Protocol
Description: Defined as completion of vaginal cuff brachytherapy followed by 3 cycles of dose dense paclitaxel and carboplatin chemotherapy
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
Participants | 27

2. Secondary Outcome: Frequency of Adverse Events Related to Acute Toxicity During Treatment
Description: Frequency and severity of adverse events as assessed by the CTCAE v4
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
Participants | 9

3. Secondary Outcome: Sites of Failure
Description: Proportion of participants who experienced failure in regional or distant sites
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
Participants | 0

4. Secondary Outcome: Recurrence-free Survival
Description: time from study entry to the first tumor recurrence
Time Frame: up to 2 years
Population: patients who received protocol therapy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
months | NA [NA to NA] — Only 3 patients recurred on study, therefore median recurrence free survival cannot be calculated.

5. Secondary Outcome: Contributing Cause of Death
Description: The contributing cause of death for patients with high risk endometrial cancer
Time Frame: up to 2 years
Population: Number of patients who died following protocol treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
Participants
  Unknown cause of death | 1
  Alive | 31

6. Secondary Outcome: Overall Survival
Description: time from study entry to death
Time Frame: up to 2 years
Population: Patients who received protocol treatment
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
Number analyzed (Participants) | 32
months | NA [NA to NA] — Only 1 patient died on study, OS cannot be calculated

ADVERSE EVENTS:
Time Frame: Deaths were assessed for up to 2 years. Adverse events were assessed for up to 4 months.
Arm/Group | Vaginal Cuff Brachytherapy + Chemotherapy
All-Cause Mortality (participants affected / at risk) | 1/32
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 10/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaginal Cuff Brachytherapy + Chemotherapy (N=32)
Fatigue (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Taxol Reaction (Immune system disorders) | 3
Anemia (Blood and lymphatic system disorders) | 2
Peripheral Neuropathy (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/46/NCT03189446/Prot_SAP_002.pdf
  • Informed Consent Form (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT03189446/ICF_003.pdf